CLINICAL TRIAL: NCT06993155
Title: A Randomized, Placebo-controlled, Double-blind, Parallel-group, Dose-response Trial Evaluating the Efficacy and Safety of Leflutrozole on Testicular Function
Brief Title: A Clinical Trial Evaluating the Efficacy and Safety of Leflutrozole on Testicular Function
Acronym: ETNA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ReproNovo Aps (Industry)
Responsible Party: Sponsor
Organization: ReproNovo SA (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RPN-LFT01
Record Dates: First submitted 2025-05-19; First posted 2025-05-28 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Semen Quality
MeSH Terms: interventions — leflutrozole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Leflutrozole, 0.05 mg (Experimental): Leflutrozole, 0.05 mg, oral capsule, once weekly for 16 weeks
  Interventions: Drug: Leflutrozole, Dose 1
- Leflutrozole, 0.1 mg (Experimental): Leflutrozole, 0.1 mg, oral capsule, once weekly for 16 weeks
  Interventions: Drug: Leflutrozole, Dose 2
- Leflutrozole, 0.3 mg (Experimental): Leflutrozole, 0.3 mg, oral capsule, once weekly for 16 weeks
  Interventions: Drug: Leflutrozole, Dose 3
- Placebo (Placebo Comparator): Placebo, oral capsule, once weekly for 16 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Leflutrozole, Dose 1 — Leflutrozole, Dose 1 once weekly for 16 weeks
  Arms: Leflutrozole, 0.05 mg
Drug: Leflutrozole, Dose 2 — Leflutrozole, Dose 2 once weekly for 16 weeks
  Arms: Leflutrozole, 0.1 mg
Drug: Leflutrozole, Dose 3 — Leflutrozole, Dose 3 once weekly for 16 weeks
  Arms: Leflutrozole, 0.3 mg
Drug: Placebo — Placebo once weekly for 16 weeks
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate three doses of the drug leflutrozole on improvement of semen quality in men. It will also study the safety of leflutrozole.

The main questions it aims to answer are:

* Does leflutrozole improve semen quality?
* What medical problems do participants experience when taking leflutrozole?

Researchers will compare leflutrozole to a placebo (a look-alike substance that contains no drug).

Participants will:

* Take leflutrozole or a placebo orally once a week for 16 weeks.
* Visit the clinic every 4 weeks for checkups and tests.
* Provide semen samples to measure changes in semen quality.
* Have their blood tested to measure hormone levels and ensure safety.
* Be monitored for any side effects.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form prior to any-related trial activity.
* Adult men aged 18-49 years (both inclusive).
* Low serum total testosterone concentration on two occasions.
* Serum Sex Hormone Binding Globulin within or above normal range at screening.
* Serum estradiol (E2) level within or above normal range at screening.
* Serum Luteinizing Hormone level within or below normal range at screening.
* Low total motile sperm count in two samples.
* Semen volume ≥1.0 mL in two samples.
* Ability to understand and comply with the requirements of the protocol.

Exclusion Criteria:

* Anatomical abnormalities of the testes or malignant or benign tumors of the testes.
* Pituitary or hypothalamic disease.
* Prostate disease.
* Treatment with one or more of the following prescription drugs or over-the-counter medications or supplements for 6 months prior to the screening visit:

  1. Compounds with androgenic or estrogenic properties (i.e., agonist or antagonist) or that affect production of sex hormones.
  2. 5-α reductase inhibitors, e.g., finasteride and dutasteride.
  3. Fertility drugs, including clomiphene, FSH, hMG and hCG preparations.
  4. Growth hormone.
  5. Opioid-receptor antagonists, e.g., naloxone and long-acting opioids.
  6. Selective α-adrenergic-receptor antagonists (alpha blockers).
  7. Topical or systemic testosterone replacement therapy (TRT).
  8. Anabolic steroids.
* Inability to reliably produce the required semen samples for trial assessments due to significant erectile dysfunction, anorgasmia, or other reasons.
* Participation in any clinical trial using clinical intervention within 3 months before the screening visit or 5 half-lives of investigational product administration, whichever is shorter.
* Any clinically significant 12-lead ECG abnormalities at screening.
* Known history of thromboembolic disease.
* Grade 3 lower extremity edema.
* Known cardiovascular disease.
* Known history of osteoporosis or fragility fractures.
* Known moderate or severe impairment of renal or hepatic function.
* Untreated diagnosis of sleep apnea.
* History of cancer within the last 5 years.
* Known alcohol and/or drug abuse within the last 12 months prior to randomization or evidence of such abuse indicated by the laboratory results during the screening assessments.
* Known chronic opioid use and/or misuse within the last 12 months prior to randomization.
* Any psychiatric or medical disorder or circumstance, which in the investigator's opinion might jeopardize participant's safety or compliance with the protocol.
* Hypersensitivity to any active ingredients or excipients in the medicinal products used in this trial.

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change in total motile sperm count (TMSC) after 16 weeks of treatment. | From baseline to the end of treatment at 16 weeks.
  Total motile sperm count will be assessed through semen analysis conducted at specialized andrology laboratories.

SECONDARY OUTCOMES:
Changes in total sperm count (TSC), sperm concentration, sperm motility, normal sperm morphology, and semen volume after 16 weeks of treatment. | From baseline to the end of treatment at 16 weeks.
  Sperm parameters will be assessed through semen analysis conducted at specialized andrology laboratories.
Percentage of participants with TMSC ≥5 million, ≥10 million, and ≥20 million after 16 weeks of treatment. | At end of treatment at 16 weeks.
  Total motile sperm count will be assessed through semen analysis conducted at specialized andrology laboratories.
Percentage of participants with a relative increase of ≥50%, ≥75% and ≥100% in TMSC after 16 weeks of treatment. | From baseline to the end of treatment at 16 weeks.
  Total motile sperm count will be assessed through semen analysis conducted at specialized andrology laboratories.
Percentage of participants with sperm DNA fragmentation index (DFI) <15%, <25% and <30% after 16 weeks of treatment. | At end of treatment at 16 weeks.
  DNA fragmentation index will be analyzed at a specialized andrology laboratory.
Percentage of participants with serum total testosterone levels within the range of 450-1000 ng/dL after 4, 8, 12 and 16 weeks of treatment. | At 4 , 8, 12 and 16 weeks of treatment.
  Blood samples will be analyzed at a central laboratory.
Percentage of participants with serum total testosterone levels within the normal range of 300-1000 ng/dL after 4, 8, 12 and 16 weeks of treatment (for participants with baseline levels <300 ng/dL). | At 4 , 8, 12 and 16 weeks of treatment.
  Blood samples will be analyzed at a central laboratory.
Changes in serum concentrations of total testosterone, free testosterone, bioavailable testosterone, SHBG, FSH, LH, estradiol, inhibin B, and total testosterone / estradiol ratio after 4, 8, 12 and 16 weeks of treatment. | From baseline to 4 , 8, 12 and 16 weeks of treatment.
  Blood samples will be analyzed at a central laboratory.
Plasma concentrations of leflutrozole after 4, 8, 12 and 16 weeks of treatment. | At 4 , 8, 12 and 16 weeks of treatment.
  Blood samples will be analyzed at a central laboratory.
Semen concentrations of leflutrozole after 12 weeks of treatment. | After 12 weeks of treatment.
  Semen analysis will be performed at a central laboratory.
Changes in libido based upon questionnaire after 4 and 16 weeks of treatment. | From baseline to 4 and 16 weeks of treatment.
  Participants will complete the Hypogonadism Impact of Symptoms Questionnaire Short Form (HIS-Q SF). The questions on libido use a 5-point scale, ranging from "never" (worst outcome) to "always" (best outcome).
Changes in energy based upon questionnaire after 4 and 16 weeks of treatment. | From baseline to 4 and 16 weeks of treatment.
  Participants will complete the Hypogonadism Impact of Symptoms Questionnaire Short Form (HIS-Q SF). The questions on energy use a 5-point scale, ranging from "not at all" (best outcome) to "extremely" (worst outcome).
Percentage of participants who overshoot testosterone at any time during the trial. | At any time during the trial
  Blood samples will be analyzed at a central laboratory
Frequency and intensity of adverse events, including serious adverse events and adverse events leading to discontinuation. | From informed consent to end of trial
  Adverse events will be collected from participant sign informed consent to end of trial
Changes in circulating levels of clinical chemistry and hematology parameters after 4, 8, 12 and 16 weeks of treatment. | From baseline to 4 , 8, 12 and 16 weeks of treatment.
  Blood samples will be analyzed at a central laboratory.
Changes in serum prostate-specific antigen (PSA) levels after 4, 8, 12 and 16 weeks of treatment. | From baseline to 4 , 8, 12 and 16 weeks of treatment.
  Blood samples will be analyzed at a central laboratory.
Changes in ECG parameters after 16 weeks of treatment. | From baseline to the end of treatment at 16 weeks.
  ECG will be measured at the trial sites and analyzed centrally.
Changes in systolic and diastolic arterial blood pressure | From baseline to 4 , 8, 12 and 16 weeks of treatment.
  Blood pressure will be taken at the trial sites.
Proportion of participants with systolic blood pressure >140 mmHg and diastolic pressure >90 mmHg | From baseline to 4 , 8, 12 and 16 weeks of treatment.
  Blood pressure will be taken at the trial sites.
Proportion of participants with systolic blood pressure >160 mmHg and diastolic pressure >110 mmHg | From baseline to 4 , 8, 12 and 16 weeks of treatment.
  Blood pressure will be taken at the trial sites.
Changes in lipids and in carbohydrate metabolism parameters after 16 weeks of treatment | From baseline to the end of treatment at 16 weeks.
  Blood samples will be analyzed at a central laboratory.
Changes in serum C-terminal cross-linking telopeptide of type 1 collagen (s-CTx) and serum procollagen type 1 N propeptide (s PINP) after 16 weeks of treatment. | From baseline to the end of treatment at 16 weeks.
  Blood samples will be analyzed at a central laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — ReproNovo Aps
Locations (4):
- United States (4):
  - ReproNovo Investigational Site, North Hollywood, California
  - ReproNovo Investigational Site, Pomona, California
  - ReproNovo Investigational Site, Garden City, New York
  - ReproNovo Investigational Site, Middleburg Heights, Ohio

IPD SHARING:
Plan to Share IPD: No